CLINICAL TRIAL: NCT00000451
Title: Naltrexone and SSRI Therapy for Alcohol Dependence in Alaska Natives
Brief Title: Drug Therapy for Alcohol Dependence in Alaska Natives (Naltrexone/Sertraline)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIAAAOMA12028; R01AA012028 (NIH)
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Alcoholism; Alcohol Dependence
Keywords: Alcoholism; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Sertraline; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Experimental): Naltrexone plus Sertraline
  Interventions: Drug: naltrexone
- 2 (Experimental): Naltrexone alone
  Interventions: Drug: sertraline; Drug: naltrexone

INTERVENTIONS:
Drug: sertraline — 16 week outpatient study
  Other Names: Zoloft
  Arms: 2
Drug: naltrexone — 16 week outpatient study
  Other Names: Revia

SUMMARY:
This study will assess the ability of naltrexone (Revia) to reduce the risk of relapse in Alaska natives with alcohol dependence. The study will also examine whether a combination of naltrexone and sertraline (Zoloft) yields better abstinence rates than naltrexone used alone. Alaska Native individuals will be recruited into a 16 week outpatient study.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native having biological Alaska Native ancestry.
* Meets criteria for alcohol dependence.
* Prior to entering the study must be abstinent between 3 and 14 days and have a withdrawal assessment.
* Stable residence to ensure that subjects can be located during the study.

Exclusion Criteria:

* Currently meets criteria for abuse or dependence on substances other than alcohol or nicotine.
* Current use of disulfiram.
* Psychotic or otherwise severely psychiatrically disabled.
* Use of other psychotropic medications including antidepressants and anxiolytics.
* Medical conditions that would not permit the use of sertraline or naltrexone, such as a history of unstable or severe hepatic, cardiovascular, metabolic, endocrine, gastrointestinal or kidney disease.
* Hepatocellular disease or elevated bilirubin levels.
* Females who are pregnant, nursing, or not using a reliable method of birth control.
* Probation or parole requirements that might interfere with participation in the study.
* Involvement in alcohol treatment other than provided by the study or AA.
* Use of monoamine oxidase inhibitors in the past month.
* Current use of Type 1C antiarrhythmics propafenone and flecainide.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2003-01; Primary Completion 2005-08 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Days abstinent

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Stephanie O'Malley, Principal Investigator — Yale University
Locations (1):
- New Haven, Connecticut, United States